CLINICAL TRIAL: NCT03445767
Title: Structured Polypharmacy Management Before Elective Non-cardiac Surgery in Frail and Elderly People: a Pilot for a Randomized Control Trial
Brief Title: Structured Polypharmacy Management Before Elective Non-cardiac Surgery in Frail and Elderly People
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive full funding to proceed
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20170663
Record Dates: First submitted 2018-01-30; First posted 2018-02-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Polypharmacy
Keywords: Peri-operative care; Medication management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): All patients will receive perioperative care per the standards of TOH. Standard care relevant to our study consists of a history by a nurse or physician; a best possible medication history performed by a pharmacy technician; and standardized perioperative-specific medication recommendations (e.g., anticoagulant, diabetes agent, and ACE-inhibitor management) based on medical directives. Medication recommendations beyond these medical directives do not occur as standard care in our clinics. Participants will be informed that their medical care will proceed as usual and that they are being recruited for a study to evaluate medication recommendations before surgery
- Intervention (Experimental): In addition to standard care, the intervention will include a structured preoperative polypharmacy management strategy that consists of: a) input of best possible medication history and comorbidities into our polypharmacy management tool (MedSafer); b) communication of the prioritized deprescribing plan (if indicated) to the patient's active treating physicians (automatically via fax), to the perioperative team (surgeon, anesthesiologist), and to the electronic medical record. During the pre-operative visit, the patient will receive a generalized information flyer about deprescribing. As in the usual care phase, patients will continue to receive usual recommendations from the perioperative team based on medical directives relevant to the perioperative period.
  Interventions: Other: MedSafer

INTERVENTIONS:
Other: MedSafer — An electronic deprescribing intervention that identifies potentially inappropriate medications (PIMs) and generates instructions for safe discontinuation. These recommendations are presented to the treating physicians for their consideration.
  Arms: Intervention

SUMMARY:
The older segment of the population is growing faster than any other segment. Older people have surgery more often than any other age group, and these older patients often take multiple medications, including medications that may result in more side effects (and risk) than benefit. Older patients who take multiple medications, and especially high risk medication, are more likely to die after surgery, and in those who survive, levels of disability are higher. For these reasons, testing a program that reviews the medications of older patients before surgery to decrease the use of dangerous medicines is very important.

Most older patients in Ontario are seen in a preoperative anesthesiology clinic. Previous research has shown that this clinic visit is a "teachable moment", where patients are more motivated to change their health-related behaviors. Therefore, the investigators propose to compare a structured medication review in the preoperative clinic to the usual care that people receive with the goal of decreasing the number and potential danger of the medications taken by older surgical patients. Recent systematic reviews have shown that no such programs have been tested to date in patients having surgery, so our findings will be unique. In addition, the investigators will also measure the impact of this program on people's health status, disability status, and use of healthcare resources (such as days in hospital) after surgery. If the investigators find that this single-center pilot randomized controlled designed study positively impacts these patient health outcomes, the investigators will perform a future multi-center cluster randomized trial of our intervention.

MedSafer is a CIHR-funded Canadian software product that aids patients and physicians in deprescribing. It contains rules that identify potentially inappropriate medications (PIMs), prioritizes them in terms of risk of harm, and provides deprescribing opportunities for safely stopping medications using the current evidence as well as incorporating patient comorbidities in the analyses.

DETAILED DESCRIPTION:
The population is aging rapidly, and elderly people have surgery at a higher rate than any other age group. Advanced age is independently associated with a 2- to 4-fold increase in adverse event rates after surgery, as well as increased rates of postoperative healthcare resource use such as costs and prolonged hospital length of stay. Polypharmacy (defined by the World Health Organization as taking >5 medications concurrently), and potentially inappropriate medications (PIM; i.e., taking medications that are likely to produce more harm than benefit given an individual's risk profile) are increasingly common in older people.

In the perioperative setting, the epidemiology of polypharmacy and inappropriate prescribing is poorly described. Single center studies of general surgery patients suggest that inappropriate prescriptions are independently associated with a 3- to 4- fold increase in the odds of serious complications, while hip fracture patients with polypharmacy have an increased risk of readmission and are often discharged on the same PIMs which may have caused the fracture.

Strategies to address polypharmacy and medication appropriateness have been synthesized in two recent systematic reviews. In general, interventions resulted in decreases in the number of medications taken, and overall medication appropriateness. However, substantial gaps in this knowledge base were also identified. First, no perioperative interventions were identified. Second, overall methodological quality of identified studies was low to very low, with significant issues identified related to study design and inadequate power, poor allocation concealment, and lack of appropriate analytic techniques. Finally, although decreasing the number and inappropriateness of medications are worthwhile outcomes, most studies did not report the impact of these interventions on patient-centered or system-level outcomes.

The preoperative anesthesiology clinic encounter may represent an optimal time to initiate polypharmacy management strategies, as the surgical encounter with the healthcare team is a teachable moment where patients demonstrate extra motivation to make positive changes in their health behaviors. Therefore, the hypothesized positive impact of preoperative polypharmacy management could extend not only into the postoperative period, but also on a longitudinal basis beyond the transition from acute postoperative care.

The preoperative polypharmacy management intervention will be based on a pragmatic, evidence-based, CIHR-funded tool developed by our coinvestigators from McGill for use in elderly inpatients. It has recently been field tested in a 600-patient inpatient study at the Universities of Ottawa, Toronto, and McGill. The tool is a web-based platform developed by experts in internal and geriatric medicine and is based on best-practice guidelines, Choosing Wisely Canada's declarative statements, and evolving issues (such as narcotic and benzodiazepine co-administration). It contains rules that identify PIMs, prioritizes them in terms of risk of harm, and provides deprescribing opportunities for safely stopping medications using the current evidence as well as incorporating patient comorbidities in the analyses.

The investigators will address a clear knowledge gap in the literature by conducting a single center pilot randomized trial to evaluate the efficacy of a structured polypharmacy management program in preparation for a future multicenter randomized trial. The primary objectives of this pilot study are to: (1) provide evidence of efficacy of the intervention in reducing PIMs, (2) estimate characteristics of secondary outcomes, specifically patient-centered and system-level measures, including baseline prevalence and measures of variation, to inform sample size calculations for a future multi-site randomized trial powered to meaningfully impact these outcomes, and (3) demonstrate acceptability of the intervention to patients and providers along with potential barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* English or French-speaking people aged 65 years or older seen in the Pre-Admission Unit prior to elective, inpatient non-cardiac surgery

Exclusion Criteria:

* Patients who cannot be reached by telephone for follow up, or are not covered by the Ontario Health Insurance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Average number of PIMs | 90-days post-surgery
  Average number of Potentially Inappropriate Medications based on patient report

SECONDARY OUTCOMES:
Patient-reported health outcomes: Health related quality of life | Before surgery, 30-day post-surgery, and 90-day post-surgery
  Standardized instrument (5 level version) developed by the EuroQol Group as a measure of health-related quality of life (patient-reported). The EQ-5D assesses domains of self-perceived mobility, self-care, usual activity participation, pain/discomfort, and anxiety depression which is captured as a overall health state score. The EQ-5D also uses a self-report 0-100 point scale relating the person's current health status to their best imaginable status.
Patient-reported health outcomes: Sleep Quality | Before surgery, 30-days post-surgery, and 90-days post-surgery
  Sleep quality measured using the PROMIS (Patient-Reported Outcomes Measurement Information System) short form 4a questions.
Patient-reported health outcomes: Disability | Before surgery, 30-days post-surgery, and 90-days post-surgery
  Disability measured using the World Health Organization Disability Assessment Schedule version 2.0, a 30-day look-back multidimensional disability scale that is validated in a variety of disease states, including postoperatively.
Adverse Events | Through study completion, an average of 7 days
  Including falls, and surgical complications using the Post-Operative Morbidity Survey which looks at several categories of complications (pulmonary, cardiovascular, neurological, gastro-intestinal, infectious, renal, wound, hematological, and pain)
Hospital length of stay | Within 365 days after surgery
  Number of days in hospital post-operatively- based on validated administrative data
Proportion of patients discharged to an institution, readmissions within 30 days of discharge | Within 365 days after surgery
  Number of patients discharged to an institution and/or re-admitted post-operatively
Patient safety indicators | Within 365 days after surgery
  A health system outcome- based on validated administrative data
Costs of hospitalization | Within 365 days after surgery
  Amount of healthcare dollars spent will be generated using a validated algorithm in our administrative data

OTHER OUTCOMES:
Feasibility outcomes: Recruitment rate | Through study completion, an average of 1 year
  Percentage of eligible patients enrolled into the study (The feasibility target is at 11 patients per month(~20% of eligible patients successfully recruited)
Feasibility outcomes: Retention Rate | Through study completion, an average of 1 year
  Percentage of patients retained for follow-up at 90-days (target of >90%)
Acceptability of the intervention to patients | Through study completion, an average of 1 year
  Patient acceptability of the application will be assessed using a 5-point likert scale based on how easy it was to use (1 being the easiest and 5 being the hardest) and if they would be willing to use the application again in the future (1 being extremely willing and 5 being extremely unwilling).
Acceptability of the intervention to providers | Through study completion, an average of 1 year
  Acceptability measured through a modified version of a validated tool (Ottawa Acceptability of decision rules instrument). The tool assesses acceptability of items including usefulness, ease of use, and efficacy for patients using a scale from strongly disagree to strongly agree, or no opinion.

IPD SHARING:
Plan to Share IPD: No